CLINICAL TRIAL: NCT02109770
Title: Development of Non-invasive Prenatal Test for Microdeletion/Duplication and Other Genetic Syndromes Based on Fetal DNA Isolated From Maternal Blood
Brief Title: Development of Non-invasive Prenatal Test for Microdeletion and Other Genetic Syndromes Based on Cell Free DNA
Acronym: Microdel Triad
Status: Completed | Type: Observational
Sponsor: Natera, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: GSN014
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Microdeletion Syndromes; Trisomy 21; Trisomy 18; Trisomy 13; Sex Chromosome Abnormalities
Keywords: 22q; DiGeorge; Angelman; Cri du chat; Miller Dieker; 1p36; Phelan McDermid; Prader Willi; Wolf Hirschorn; Smith Magenis; Trisomy 21; Down syndrome; Trisomy 18; Edwards syndrome; Trisomy 13; Patau syndrome; Monosomy X; Turner syndrome; XXY; Klinefelter syndrome; XXX; XYY
MeSH Terms: conditions — Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome; Sex Chromosome Aberrations; Turner Syndrome; Klinefelter Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Maternal blood sample
  * Affected child blood sample
  * Unaffected sibling blood sample
  * Father buccal or blood sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mother child diads or triads: Families with child affected by genetic anomaly, microdeletion, microduplication, or chromosomal anomaly

SUMMARY:
The purpose of this study is to collect blood from families with a child who has been diagnosed with a chromosomal disorder including microdeletions in order to further develop a non-invasive prenatal screening test based on fetal DNA isolated from maternal blood.

DETAILED DESCRIPTION:
The primary purpose of this study is to collect family triads from families affected by a genetic or microdeletion/duplication (MD/D) syndrome to further develop non-invasive prenatal testing based on fetal DNA isolated from maternal blood. To assist with the development of the test, we will need to collect blood samples from women whose child was diagnosed with a genetic or MD/D syndrome, a blood sample from that child as well as a blood sample from their confirmed unaffected siblings. Since the test is based on Natera's Parental Support™ technology, buccal or blood samples from the biological fathers will also be requested.

A recent abstract from a five year study on prenatal microarray testing revealed that 1.6% of women who present for routine prenatal indications have a positive microarray test. With the frequency of microdeletions and microduplications (MD/D) now known to be higher than previously thought, the field is likely to move toward offering invasive testing for microarray abnormalities to all pregnant women. Although non-invasive prenatal testing for aneuploidy is now clinically available, it has become clear that non-invasive prenatal testing for MD/D is equally important. However, access to these samples is made difficult as the standard of care for offering microarray analysis to all pregnant women will take time to come to fruition. We would like to develop this non-invasive as the standard of care so that less women will have to undergo invasive testing for the diagnosis of microarray abnormalities. Thus, there is an unmet need for the development of novel tests that would increase the scope of non-invasive prenatal screening.

ELIGIBILITY:
Inclusion Criteria:

* Couples who have a child diagnosed with an autosomal chromosome abnormality (e.g. Down syndrome, Edwards syndrome, Patau syndrome).
* Couples who have a child diagnosed with a sex chromosome abnormality (e.g. Turner syndrome, Klinefelter syndrome, Triple X syndrome, 47, XYY).
* Couples who have a child diagnosed with a microdeletion/duplication syndrome (a positive microarray test).

Exclusion criteria:

* Not an English language or Spanish language speaker
* Genetics report is not available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Families with a child affected by a chromosomal abnormality.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity and Specificity of the test to diagnose chromosomal microdeletions and aneuploidy in a fetus | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Kim Martin, MD, Principal Investigator — Natera, Inc.
Locations (2):
- United States (2):
  - Natera, San Carlos, California
  - Children's Hospital Of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Wapner RJ, Babiarz JE, Levy B, Stosic M, Zimmermann B, Sigurjonsson S, Wayham N, Ryan A, Banjevic M, Lacroute P, Hu J, Hall MP, Demko Z, Siddiqui A, Rabinowitz M, Gross SJ, Hill M, Benn P. Expanding the scope of noninvasive prenatal testing: detection of fetal microdeletion syndromes. Am J Obstet Gynecol. 2015 Mar;212(3):332.e1-9. doi: 10.1016/j.ajog.2014.11.041. Epub 2014 Dec 2. PMID 25479548